CLINICAL TRIAL: NCT06773052
Title: The Experience, Perceptions and Unexpressed Needs of Heart and Lung Transplant Patients Admitted to Intensive Care: a Qualitative, Descriptive Phenomenological Observational Study
Brief Title: The Experience, Perceptions and Unexpressed Needs of Heart and Lung Transplant Patients Admitted to Intensive Care
Acronym: ReF2201
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ReF2201
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Heart and Lung Transplants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Qualitative descriptive phenomenological study aimed to investigate the experience, perceptions and unexpressed needs of patients undergoing heart and lung transplantation admitted to intensive care unit through semi-structured interviews

DETAILED DESCRIPTION:
It was conduct a qualitative phenomenological study which, through semi-structured interviews to investigate the experience , the perceptions and the unexpressed needs of patients undergoing heart and lung transplants within the specific context of " High Intensity Cardio-Thoraco-Vascular Hospitalization" of the IRCCS University Hospital of Bologna. The study aims at helping nurses to provide more adequate care, in order to meet the individual needs of patients and describe the meaning and essence of the hospitalization experience, through the in-depth analysis of the specific words pronounced by the patients themselves.

Below are the questions that guided the research:

What is the general experience of the intensive care patients? What are the experiences, the perceptions and the unexpressed needs of these patients in relation to their hospitalization in intensive care?

ELIGIBILITY:
Inclusion Criteria:

* able to understand and communicate in Italian
* transferred from intensive to sub-intensive care unit
* not affected by cognitive disorders
* who provides informed consent to the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The total sample consisted of 21 patients who underwent heart or lung transplants. Of these, 18 patients (86%) had undergone heart transplants, while 3 patients (14%) had undergone lung transplants.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Experience, perceptions and unexpressed needs of heart and lung transplant patients | through study completion, an average of 1 year
  This is a prospective qualitative descriptive observational study. Each enrolled patient will undergo a single semi-structured interview.
  Following the semi-structured interview technique, the Investigator will have a list of questions to guide the interview and to remains topic-centered. The questions are open-ended.
  The questionnaire will be structured into two macro areas:
  Questions related to the general experience of the ICU patient; Questions related to the experiences, perceptions and unexpressed needs of ICU patients (including personal impressions of hospital staff).
  To avoid potential conditioning and to promote the free expression of the subjects, the interviews will be conducted by a Investigator who is part of ICU research team but not directly involved in patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Nikita Valentina Ugenti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

REFERENCES:
- [Derived] Ugenti NV, Quirini S, Aleandri M, Di Filippo V, Durante S, Ferretti A, Guerrieri C, Martella C, Peghetti A, Sgarzi S, Valentini S, Vetromile A, Lia E. Experiences, perceptions and unexpressed needs of patients undergoing heart and lung transplantation in intensive care unit: a qualitative phenomenological study. Front Psychol. 2025 Sep 9;16:1646086. doi: 10.3389/fpsyg.2025.1646086. eCollection 2025. PMID 40994850